CLINICAL TRIAL: NCT02157805
Title: Effect of Technological Processes on Nutritional Quality of Meat Proteins
Brief Title: Technological Processes on Quality of Meat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government)
Responsible Party: Principal Investigator, Yves Boirie, PU-PH, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AU1024; 2013-A00020-45 (Registry Identifier: IDRCB number)
Record Dates: First submitted 2014-01-14; First posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Sarcopenia
Keywords: Meat processes; Amino acids bioavailability; Digestion rate; Protein synthesis; Aging; Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Red Meat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rare beef meat (Active Comparator): beef meat cooked during 5 minutes at 55°C
  Interventions: Other: beef meat
- well cook beef meat (Active Comparator): beef meat cooked during 30 minutes à 90°C
  Interventions: Other: beef meat

INTERVENTIONS:
Other: beef meat — Meat cooking conditions
  1. st condition : beef meat cooked during 5 minutes at 55°C
  2. nd condition : beef meat cooked during 30 minutes à 90°C

SUMMARY:
This project aims to assess the impact of technological processes of meat, as cooking conditions, on amino acid bioavailability and protein metabolism. The hypothesis is that, even if meat is considered as a good provider of fast proteins and so could be useful to prevent sarcopenia in aged people, the manner it is cooked can change its digestion rate and amino acids bioavailability for muscle synthesis.

DETAILED DESCRIPTION:
Beef meat, whose proteins were intrinsically labelled with 15 N, was previously obtained by infusing 15N ammonium sulphate during 50 days in the rumen of an heifer. Two different cooking conditions have been applied to this meat (5 min at 55°C vs 30 min at 90°C). Ten healthy elderly volunteers will test each processed meat according to a cross-over design, during 2 different metabolic studies separated by at least 2 weeks. Volunteers will be submitted to a diet controlled for its protein content, for 4 days (1.2 g protein/kg/day) before each metabolic investigation.

On the 2 days of metabolic investigations, after an overnight fast, blood samples will be collected for basal measurements. Then the subjects will be perfused with L-[1-13C] leucine for 9h30 hours, during which expired gas and blood samples will be regularly taken, and CO2 production measured. The volunteers will be asked to eat a 130 g beef meat 2.5h after the onset of the perfusion. Isotopic enrichments in expired gas, in plasma alpha-cetoiscaproate and in free leucine will be measured to determine whole body amino acids fluxes (oxidation, protein synthesis and proteolysis). 15N enrichments of leucine will allow splanchnic extraction measurement.

ELIGIBILITY:
Inclusion Criteria :

* Male
* Age > 70
* Body mass index 21 < BMI < 28 kg/m2
* Affiliated to National Health Insurance
* Subject giving his written informed consent
* Subject considered as normal after clinical and medical examinations

Exclusion Criteria :

* Positive serologies to HIV or HCV, or abnormal laboratory tests
* Previous medical and/or surgery judged by the investigator as incompatible with this study
* Person who doesn't eat beef or only if prepared according to religious rite
* Person wearing a removable denture or suffering of dry mouth syndrome
* Regular medication with glucocorticoids
* Intense sports activity > 7h/week
* Heavy alcohol consumption
* Being under someone's supervision
* Refusal to be registered on the National Volunteers Data file
* Being in exclusion on the National Volunteers Data file

Min Age: 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Plasma amino acids concentrations before and during 7 hours after eating labelled meat. | up to 7 hours
  Plasma amino acids concentrations before and during 7 hours after eating labelled meat.
  Splanchnic extraction of leucine. Isotopic enrichments in expired gas, in plasma alpha-cetoisocaproate and in free leucine to determine whole body protein metabolism

SECONDARY OUTCOMES:
Changes in plasma peptidome after ingestion of a meat meal | up to 7 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yves Boirie, Md-PhD, Principal Investigator — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- Centre de Recherche en Nutrition Humaine, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Derived] Buffiere C, Gaudichon C, Hafnaoui N, Migne C, Scislowsky V, Khodorova N, Mosoni L, Blot A, Boirie Y, Dardevet D, Sante-Lhoutellier V, Remond D. In the elderly, meat protein assimilation from rare meat is lower than that from meat that is well done. Am J Clin Nutr. 2017 Nov;106(5):1257-1266. doi: 10.3945/ajcn.117.158113. Epub 2017 Sep 13. PMID 28903955